CLINICAL TRIAL: NCT03286231
Title: Anti-FLEX: Flexed Levering of Gluteal Vessels on OR Table May Lead to Extreme Danger During Gluteal Augmentation With Lipoaspirate, a Radio-graphically Studied Position of Superior and Inferior Gluteal Vessels During Flexion of OR Table or "Jack-knife" Position, Danger Zone.
Brief Title: Anti-FLEX: Flexed Levering of Gluteal Vessels
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00031729
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Healthy
Keywords: gluteal venous vasculature; prone position; jackknife position
MeSH Terms: interventions — Postmortem Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy volunteers: Healthy volunteers who will undergo contrast-enhanced CT imaging of the gluteal venous vasculature in the prone and jackknife positions
  Interventions: Diagnostic Test: CT imaging

INTERVENTIONS:
Diagnostic Test: CT imaging — Contrast-enhanced CT imaging of the pelvis in prone and jackknife positions

SUMMARY:
The purpose of this study is to evaluate the effect of the gluteal vasculature in the prone and jackknife positions.

DETAILED DESCRIPTION:
This is a prospective collection of contrast-enhanced CT images of healthy female volunteers in prone and jackknife positions in order to determine if position impacts gluteal venous vasculature.

ELIGIBILITY:
Inclusion Criteria:

* Females age 20 - 50 years
* BMI between 20 - 35 kg/m2
* Willingness and ability to provide written informed consent
* Willingness and ability to comply with all study procedures
* Interested or planning to have a gluteal augmentation

Exclusion Criteria:

* Males
* Females age < 20 or >= 51 years
* BMI between < 20 or > 35 kg/m2
* Prior gluteal augmentation surgery
* Any prior gluteal soft tissue filler
* Known or suspected history of immediate or delayed hypersensitivity (including but not limited to hives, anaphylactoid or cardiovascular reactions, laryngeal edema, and bronchospasm) to iodine or any iodinated contrast medium
* Documented history of chronic kidney disease that contraindicates the use of contrast dye
* Pregnant
* Currently breast-feeding
* Any reason (in addition to those listed above) that, in the opinion of the principal investigator, precludes full participation in the study

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females only
Study Population: Healthy volunteers who will undergo contrast-enhanced CT imaging of the gluteal venous vasculature in the prone and jackknife positions
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
Mean difference of position of the gluteal venous vasculature in relation to the skin | at CT scan visit
  Between the Prone position and the Jackknife position

SECONDARY OUTCOMES:
Mean difference of vessel diameter of the gluteal venous vasculature | at CT scan visit
  Between the Prone position and the Jackknife position
Mean difference of the danger zone | at CT scan visit
  Between the Prone position and the Jackknife position

CONTACTS AND LOCATIONS:
Overall Officials: Connor Barnes, MD, Principal Investigator — University of South Florida
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Illouz YG. The fat cell "graft": a new technique to fill depressions. Plast Reconstr Surg. 1986 Jul;78(1):122-3. No abstract available. PMID 3725947
- [Background] Hsu VM, Stransky CA, Bucky LP, Percec I. Fat grafting's past, present, and future: why adipose tissue is emerging as a critical link to the advancement of regenerative medicine. Aesthet Surg J. 2012 Sep;32(7):892-9. doi: 10.1177/1090820X12455658. PMID 22942117
- [Background] Cardenas-Camarena L, Arenas-Quintana R, Robles-Cervantes JA. Buttocks fat grafting: 14 years of evolution and experience. Plast Reconstr Surg. 2011 Aug;128(2):545-555. doi: 10.1097/PRS.0b013e31821b640b. PMID 21788847
- [Background] Toledo LS. Gluteal augmentation with fat grafting: the Brazilian buttock technique: 30 years' experience. Clin Plast Surg. 2015 Apr;42(2):253-61. doi: 10.1016/j.cps.2014.12.004. PMID 25827567
- [Background] LINCOLN JR, SAWYER HP Jr. Complications related to body positions during surgical procedures. Anesthesiology. 1961 Sep-Oct;22:800-9. doi: 10.1097/00000542-196109000-00014. No abstract available. PMID 14465376
- [Background] Astarita DC, Scheinin LA, Sathyavagiswaran L. Fat transfer and fatal macroembolization. J Forensic Sci. 2015 Mar;60(2):509-10. doi: 10.1111/1556-4029.12549. Epub 2015 Feb 4. PMID 25653075
- [Result] Mofid MM, Teitelbaum S, Suissa D, Ramirez-Montanana A, Astarita DC, Mendieta C, Singer R. Report on Mortality from Gluteal Fat Grafting: Recommendations from the ASERF Task Force. Aesthet Surg J. 2017 Jul 1;37(7):796-806. doi: 10.1093/asj/sjx004. PMID 28369293
- [Result] Klein SM, Prantl L, Geis S, Eisenmann-Klein M, Dolderer J, Felthaus O, Loibl M, Heine N. Pressure monitoring during lipofilling procedures. Clin Hemorheol Microcirc. 2014;58(1):9-17. doi: 10.3233/CH-141872. PMID 25227189
- [Result] Katayama H, Yamaguchi K, Kozuka T, Takashima T, Seez P, Matsuura K. Adverse reactions to ionic and nonionic contrast media. A report from the Japanese Committee on the Safety of Contrast Media. Radiology. 1990 Jun;175(3):621-8. doi: 10.1148/radiology.175.3.2343107.